CLINICAL TRIAL: NCT04307056
Title: EVALUATION OF HIGH INTENSITY FOCUSED ULTRASOUND (HIFU) IN CURATIVE TREATMENT OF LOCALIZED PROSTATE CANCER AT LOW OR INTERMEDIATE RISK AND IN TREATMENT OF RECURRENCE AFTER RADIOTHERAPY (FORFAIT INNOVATION ART L165-1-1 Social Security Code)
Brief Title: Evaluation of HIFU in TREATMENT OF LOCALIZED PROSTATE CANCER and OF RECURRENCE AFTER RADIOTHERAPY
Acronym: HIFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Francaise d'Urologie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/AFU/12.03; 2013-A01042-43 (Other: ANSM)
Record Dates: First submitted 2020-02-07; First posted 2020-03-13 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-11

CONDITIONS: Prostate Cancer; Ultrasound Therapy
Keywords: HIFU
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFU (Experimental): Patients Treated with high intensity focused ultrasound (HIFU)
  Interventions: Procedure: High Intensity Focused Ultrasound (HIFU) Treatment
- Prostatectomy (Active Comparator): Patients Treated by Radical Prostatectomy
  Interventions: Procedure: Radical Prostatectomy

INTERVENTIONS:
Procedure: Radical Prostatectomy — The surgical approach can be open or laparoscopic. The procedure begins with lymph node dissection for the intermediate risk groups (PSA > 10 ng/mL and/or presence of grade 4 Gleason score). Total prostatectomy includes removal of the seminal vesicles. It can preserve 1 or 2 neurovascular bundles, depending on the cancer stage and/or the choice expressed by the patient. The vesicourethral suture is either a running or interrupted suture, and there is drainage by a bladder catheter for at least 5 days.
  Arms: Prostatectomy
Procedure: High Intensity Focused Ultrasound (HIFU) Treatment — The treatment with High Intensity Focused Ultrasound (HIFU) evaluated in this study will be delivered by 2 types of medical devices currently available on the market, Ablatherm® and Focal One®. They are both computer-controlled and provided with an endo-rectal probe with integrated ultrasound, enabling planning and the monitoring of treatment of localized prostate cancer in realtime.
  Arms: HIFU

SUMMARY:
to compare the efficacy of HIFU treatment with standard treatment in two situations:

1. as first-line cancer treatment, HIFU is compared to radical prostatectomy.
2. for patients with recurrence after external beam radiotherapy, HIFU treatment is compared to radical prostatectomy.

ELIGIBILITY:
General inclusion criteria

* Patients with localized adenocarcinoma of the prostate classified as T1-2, N0, Nx M0
* classified as low or intermediate risk
* Patient with PSA < 15 ng/ml, Gleason score ≤ 7 restricted to the form [3 + 4].
* Biopsy with at least 12 specimens and a maximum of four out of six invaded sextants
* Patient with a pelvic MRI if there is an intermediate risk and a bone scintigraphy if PSA > 10 ng/ml
* Patient affiliated with health insurance or beneficiary of an equivalent plan

Inclusion criteria for the HIFU Arm

* Patients 70 years of age or older
* Patients with a life expectancy related to age and associated illness estimated to be greater than 5 years

Inclusion Criteria for Total Prostatectomy Arm

• Patients with a life expectancy greater than 10 years and a state of health allowing general anaesthesia.

NON-INCLUSION CRITERIA

* Patient participating in other biomedical research within 3 months prior to their inclusion in this protocol
* Included patient simultaneously participating in another research study

Min Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3862 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival | 30 months
  The main objective for patients is to compare recurrence-free survival (i.e., the rate of salvage therapy by external beam radiotherapy and/or hormone therapy) in patients treated by HIFU and those treated by radical prostatectomy. The implementation of salvage therapy will be decided according to several non-exclusive criteria (positivity of margins (for patients with radical prostatectomy), PSA at 3 months, biologic recurrence (increase in PSA > 0.2 ng/ml after radical surgery, > Nadir +2 after HIFU), control biopsies positive, the appearance of metastases

SECONDARY OUTCOMES:
Immediate or late complications | 6 weeks after treatment
  clinical observations (Stenosis, bleeding, hemorrhoids, urinary infections ...)
Immediate or late complications | Day 0, Inclusion
  clinical observations (Stenosis, bleeding, hemorrhoids, urinary infections ...)
immediate or late complications | 3 months after treatment
  clinical observations (Stenosis, bleeding, hemorrhoids, urinary infections ...)
immediate or late complications | 6 months after treatment
  clinical observations (Stenosis, bleeding, hemorrhoids, urinary infections ...)
immediate or late complications | 12 months after treatment
  clinical observations (Stenosis, bleeding, hemorrhoids, urinary infections ...)
immediate or late complications | 18 months after treatment
  clinical observations (Stenosis, bleeding, hemorrhoids, urinary infections ...)
immediate or late complications | 24 months after treatment
  clinical observations (Stenosis, bleeding, hemorrhoids, urinary infections ...)
immediate or late complications | 30 months after treatment
  clinical observations (Stenosis, bleeding, hemorrhoids, urinary infections ...)
urinary function | Day 0, Inclusion
  measured by the International Prostate Symptom score (IPSS). For the first seven questions: 0 to 7: mild disorders, 8 to 19: moderate disorders, 20 to 35: severe disorders For quality of life question 8: Score from 0 to 6: 0 no discomfort, 6 very discomfort
urinary function | 6 months after treatment
  measured by the International Prostate Symptom score (IPSS). For the first seven questions: 0 to 7: mild disorders, 8 to 19: moderate disorders, 20 to 35: severe disorders For quality of life question 8: Score from 0 to 6: 0 no discomfort, 6 very discomfort
urinary function | 12 months after treatment
  measured by the International Prostate Symptom score (IPSS). For the first seven questions: 0 to 7: mild disorders, 8 to 19: moderate disorders, 20 to 35: severe disorders For quality of life question 8: Score from 0 to 6: 0 no discomfort, 6 very discomfort
urinary function | 24 months after treatment
  measured by the International Prostate Symptom score (IPSS). For the first seven questions: 0 to 7: mild disorders, 8 to 19: moderate disorders, 20 to 35: severe disorders For quality of life question 8: Score from 0 to 6: 0 no discomfort, 6 very discomfort
urinary function | 30 months after treatment
  measured by the International Prostate Symptom score (IPSS). For the first seven questions: 0 to 7: mild disorders, 8 to 19: moderate disorders, 20 to 35: severe disorders For quality of life question 8: Score from 0 to 6: 0 no discomfort, 6 very discomfort
urinary function | Day 0, Inclusion
  Urinary function measured by the International Continence Society score (ICS score). Question 1: Stress incontinence Score (frequency) from 0 to 4 (never - always) Sub-score 1a (quality of life) from 0 to 3 (none - significant discomfort) Question 2: Insensitive incontinence Score (frequency) from 0 to 4 (never - always) Sub score 2 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 3: Incontinence at night Score (frequency) from 0 to 4 (never - always) Sub score 3 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 4: Change of clothing or protective wear Score from 0 to 4 (no leakage of urine - seal port) Sub-score 4 bis (quality of life) from 0 to 3 (no significant discomfort to major discomfort) Question 5: Number of protection used Day Score: 0 to 4 (none to 6 or more) Score at night: 0 to 4 (none to 6 or more)
  Translated with www.DeepL.com/Translator (free version)
urinary function | 6 months after treatment
  Urinary function measured by the International Continence Society score (ICS score). Question 1: Stress incontinence Score (frequency) from 0 to 4 (never - always) Sub-score 1a (quality of life) from 0 to 3 (none - significant discomfort) Question 2: Insensitive incontinence Score (frequency) from 0 to 4 (never - always) Sub score 2 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 3: Incontinence at night Score (frequency) from 0 to 4 (never - always) Sub score 3 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 4: Change of clothing or protective wear Score from 0 to 4 (no leakage of urine - seal port) Sub-score 4 bis (quality of life) from 0 to 3 (no significant discomfort to major discomfort) Question 5: Number of protection used Day Score: 0 to 4 (none to 6 or more) Score at night: 0 to 4 (none to 6 or more)
  Translated with www.DeepL.com/Translator (free version)
urinary function | 12 months after treatment
  Urinary function measured by the International Continence Society score (ICS score). Question 1: Stress incontinence Score (frequency) from 0 to 4 (never - always) Sub-score 1a (quality of life) from 0 to 3 (none - significant discomfort) Question 2: Insensitive incontinence Score (frequency) from 0 to 4 (never - always) Sub score 2 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 3: Incontinence at night Score (frequency) from 0 to 4 (never - always) Sub score 3 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 4: Change of clothing or protective wear Score from 0 to 4 (no leakage of urine - seal port) Sub-score 4 bis (quality of life) from 0 to 3 (no significant discomfort to major discomfort) Question 5: Number of protection used Day Score: 0 to 4 (none to 6 or more) Score at night: 0 to 4 (none to 6 or more)
  Translated with www.DeepL.com/Translator (free version)
urinary function | 18 months after treatment
  Urinary function measured by the International Continence Society score (ICS score). Question 1: Stress incontinence Score (frequency) from 0 to 4 (never - always) Sub-score 1a (quality of life) from 0 to 3 (none - significant discomfort) Question 2: Insensitive incontinence Score (frequency) from 0 to 4 (never - always) Sub score 2 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 3: Incontinence at night Score (frequency) from 0 to 4 (never - always) Sub score 3 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 4: Change of clothing or protective wear Score from 0 to 4 (no leakage of urine - seal port) Sub-score 4 bis (quality of life) from 0 to 3 (no significant discomfort to major discomfort) Question 5: Number of protection used Day Score: 0 to 4 (none to 6 or more) Score at night: 0 to 4 (none to 6 or more)
  Translated with www.DeepL.com/Translator (free version)
urinary function | 24 months after treatment
  Urinary function measured by the International Continence Society score (ICS score). Question 1: Stress incontinence Score (frequency) from 0 to 4 (never - always) Sub-score 1a (quality of life) from 0 to 3 (none - significant discomfort) Question 2: Insensitive incontinence Score (frequency) from 0 to 4 (never - always) Sub score 2 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 3: Incontinence at night Score (frequency) from 0 to 4 (never - always) Sub score 3 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 4: Change of clothing or protective wear Score from 0 to 4 (no leakage of urine - seal port) Sub-score 4 bis (quality of life) from 0 to 3 (no significant discomfort to major discomfort) Question 5: Number of protection used Day Score: 0 to 4 (none to 6 or more) Score at night: 0 to 4 (none to 6 or more)
  Translated with www.DeepL.com/Translator (free version)
urinary function | 30 months after treatment
  Urinary function measured by the International Continence Society score (ICS score). Question 1: Stress incontinence Score (frequency) from 0 to 4 (never - always) Sub-score 1a (quality of life) from 0 to 3 (none - significant discomfort) Question 2: Insensitive incontinence Score (frequency) from 0 to 4 (never - always) Sub score 2 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 3: Incontinence at night Score (frequency) from 0 to 4 (never - always) Sub score 3 bis (quality of life) from 0 to 3 (none - significant discomfort) Question 4: Change of clothing or protective wear Score from 0 to 4 (no leakage of urine - seal port) Sub-score 4 bis (quality of life) from 0 to 3 (no significant discomfort to major discomfort) Question 5: Number of protection used Day Score: 0 to 4 (none to 6 or more) Score at night: 0 to 4 (none to 6 or more)
  Translated with www.DeepL.com/Translator (free version)
urinary function | Day 0, Inclusion
  Urinary function measured by the Urinary Symptom Score(USP). 3 sub-scores:
  stress urinary incontinence score: 0 to 9 (none - significant) OAB score: 0 to 21(none - significant) Dysuria score: 0 to 9 (none - significant)
urinary function | 6 months after treatment
  Urinary function measured by the Urinary Symptom Score(USP). 3 sub-scores:
  stress urinary incontinence score: 0 to 9 (none - significant) OAB score: 0 to 21(none - significant) Dysuria score: 0 to 9 (none - significant)
urinary function | 12 months after treatment
  Urinary function measured by the Urinary Symptom Score(USP). 3 sub-scores:
  stress urinary incontinence score: 0 to 9 (none - significant) OAB score: 0 to 21(none - significant) Dysuria score: 0 to 9 (none - significant)
urinary function | 18 months after treatment
  Urinary function measured by the Urinary Symptom Score(USP). 3 sub-scores:
  stress urinary incontinence score: 0 to 9 (none - significant) OAB score: 0 to 21(none - significant) Dysuria score: 0 to 9 (none - significant)
urinary function | 24 months after treatment
  Urinary function measured by the Urinary Symptom Score(USP). 3 sub-scores:
  stress urinary incontinence score: 0 to 9 (none - significant) OAB score: 0 to 21(none - significant) Dysuria score: 0 to 9 (none - significant)
urinary function | 30 months after treatment
  Urinary function measured by the Urinary Symptom Score(USP). 3 sub-scores:
  stress urinary incontinence score: 0 to 9 (none - significant) OAB score: 0 to 21(none - significant) Dysuria score: 0 to 9 (none - significant)
sexual fonction | Day 0, Inclusion
  Sexual function results are measured by the International Index Erectile Function score (IIEF-5). score from 1 to 4: not interpretable score from 5 to 10: severe erectile dysfunction score from 11 to 15: moderate erectile dysfunction score from 16 to 20: mild erectile dysfunction score from 21 to 25: normal erectile function
sexual fonction | 6 months after treatment
  Sexual function results are measured by the International Index Erectile Function score (IIEF-5). score from 1 to 4: not interpretable score from 5 to 10: severe erectile dysfunction score from 11 to 15: moderate erectile dysfunction score from 16 to 20: mild erectile dysfunction score from 21 to 25: normal erectile function
sexual fonction | 12 months after treatment
  Sexual function results are measured by the International Index Erectile Function score (IIEF-5). score from 1 to 4: not interpretable score from 5 to 10: severe erectile dysfunction score from 11 to 15: moderate erectile dysfunction score from 16 to 20: mild erectile dysfunction score from 21 to 25: normal erectile function
sexual fonction | 24 months after treatment
  Sexual function results are measured by the International Index Erectile Function score (IIEF-5). score from 1 to 4: not interpretable score from 5 to 10: severe erectile dysfunction score from 11 to 15: moderate erectile dysfunction score from 16 to 20: mild erectile dysfunction score from 21 to 25: normal erectile function
sexual fonction | 30 months after treatment
  Sexual function results are measured by the International Index Erectile Function score (IIEF-5). score from 1 to 4: not interpretable score from 5 to 10: severe erectile dysfunction score from 11 to 15: moderate erectile dysfunction score from 16 to 20: mild erectile dysfunction score from 21 to 25: normal erectile function
Evaluation of quality of life | Day 0, Inclusion
  Quality of life measured by EORTC-QLQ-C30. Questions 1 to 28 (general) score from 0 to 4 for each question (not at all to many) Question 29 (health status) score from 1 to 7 (very bad to excellent) Question 30 (quality of life) score from 1 to 7 (very bad to excellent)
Evaluation of quality of life | 6 months after treatment
  Quality of life measured by EORTC-QLQ-C30. Questions 1 to 28 (general) score from 0 to 4 for each question (not at all to many) Question 29 (health status) score from 1 to 7 (very bad to excellent) Question 30 (quality of life) score from 1 to 7 (very bad to excellent)
Evaluation of quality of life | 12 months after treatment
  Quality of life measured by EORTC-QLQ-C30. Questions 1 to 28 (general) score from 0 to 4 for each question (not at all to many) Question 29 (health status) score from 1 to 7 (very bad to excellent) Question 30 (quality of life) score from 1 to 7 (very bad to excellent)
Evaluation of quality of life | 18 months after treatment
  Quality of life measured by EORTC-QLQ-C30. Questions 1 to 28 (general) score from 0 to 4 for each question (not at all to many) Question 29 (health status) score from 1 to 7 (very bad to excellent) Question 30 (quality of life) score from 1 to 7 (very bad to excellent)
Evaluation of quality of life | 24 months after treatment
  Quality of life measured by EORTC-QLQ-C30. Questions 1 to 28 (general) score from 0 to 4 for each question (not at all to many) Question 29 (health status) score from 1 to 7 (very bad to excellent) Question 30 (quality of life) score from 1 to 7 (very bad to excellent)
Evaluation of quality of life | 30 months after treatment
  Quality of life measured by EORTC-QLQ-C30. Questions 1 to 28 (general) score from 0 to 4 for each question (not at all to many) Question 29 (health status) score from 1 to 7 (very bad to excellent) Question 30 (quality of life) score from 1 to 7 (very bad to excellent)
Evaluation of quality of life | Day 0, Inclusion
  Quality of life measured by PR 25. Questions 1 to 9 (urinary disorders) score from 0 to 4 for each question (none to many) Questions 10 to 13 (intestinal disorders) score from 0 to 4 for each question (none to many) Question 14 (hot flashes) score from 0 to 4 for each question (none to many) Question 15 (gynecomastia) score from 0 to 4 for each question (none to many) Question 16 (swollen legs) score from 0 to 4 for each question (none to many) Questions 17 to 18 (weight gain or loss) score from 0 to 4 for each question (none to many) Questions 19 to 25 (sexuality) score from 0 to 4 for each question (none to many)
Evaluation of quality of life | 6 months after treatment
  Quality of life measured by PR 25. Questions 1 to 9 (urinary disorders) score from 0 to 4 for each question (none to many) Questions 10 to 13 (intestinal disorders) score from 0 to 4 for each question (none to many) Question 14 (hot flashes) score from 0 to 4 for each question (none to many) Question 15 (gynecomastia) score from 0 to 4 for each question (none to many) Question 16 (swollen legs) score from 0 to 4 for each question (none to many) Questions 17 to 18 (weight gain or loss) score from 0 to 4 for each question (none to many) Questions 19 to 25 (sexuality) score from 0 to 4 for each question (none to many)
Evaluation of quality of life | 12 months after treatment
  Quality of life measured by PR 25. Questions 1 to 9 (urinary disorders) score from 0 to 4 for each question (none to many) Questions 10 to 13 (intestinal disorders) score from 0 to 4 for each question (none to many) Question 14 (hot flashes) score from 0 to 4 for each question (none to many) Question 15 (gynecomastia) score from 0 to 4 for each question (none to many) Question 16 (swollen legs) score from 0 to 4 for each question (none to many) Questions 17 to 18 (weight gain or loss) score from 0 to 4 for each question (none to many) Questions 19 to 25 (sexuality) score from 0 to 4 for each question (none to many)
Evaluation of quality of life | 18 months after treatment
  Quality of life measured by PR 25. Questions 1 to 9 (urinary disorders) score from 0 to 4 for each question (none to many) Questions 10 to 13 (intestinal disorders) score from 0 to 4 for each question (none to many) Question 14 (hot flashes) score from 0 to 4 for each question (none to many) Question 15 (gynecomastia) score from 0 to 4 for each question (none to many) Question 16 (swollen legs) score from 0 to 4 for each question (none to many) Questions 17 to 18 (weight gain or loss) score from 0 to 4 for each question (none to many) Questions 19 to 25 (sexuality) score from 0 to 4 for each question (none to many)
Evaluation of quality of life | 24 months after treatment
  Quality of life measured by PR 25. Questions 1 to 9 (urinary disorders) score from 0 to 4 for each question (none to many) Questions 10 to 13 (intestinal disorders) score from 0 to 4 for each question (none to many) Question 14 (hot flashes) score from 0 to 4 for each question (none to many) Question 15 (gynecomastia) score from 0 to 4 for each question (none to many) Question 16 (swollen legs) score from 0 to 4 for each question (none to many) Questions 17 to 18 (weight gain or loss) score from 0 to 4 for each question (none to many) Questions 19 to 25 (sexuality) score from 0 to 4 for each question (none to many)
Evaluation of quality of life | 30 months after treatment
  Quality of life measured by PR 25. Questions 1 to 9 (urinary disorders) score from 0 to 4 for each question (none to many) Questions 10 to 13 (intestinal disorders) score from 0 to 4 for each question (none to many) Question 14 (hot flashes) score from 0 to 4 for each question (none to many) Question 15 (gynecomastia) score from 0 to 4 for each question (none to many) Question 16 (swollen legs) score from 0 to 4 for each question (none to many) Questions 17 to 18 (weight gain or loss) score from 0 to 4 for each question (none to many) Questions 19 to 25 (sexuality) score from 0 to 4 for each question (none to many)
Evaluation of quality of life | Day 0, Inclusion
  Quality of life measured by the 3-level version of EQ-5D. Questions 1 to 3 (mobility)
  1 (no problem) to 3 (unable) Questions 4 to 6 (personal autonomy)
  1 (no problem) to 3 (unable) Questions 7 to 9 (current activities)
  1 (no problem) to 3 (unable) Questions 10 to 12 (pain/discomfort)
  1 (none) to 3 (extreme) Questions 13 to 15 (anxiety/depression)
  1 (none) to 3 (extreme) Question 16 (health status) Scale from 0 to 100 (worse health to better health)
Evaluation of quality of life | 6 months after treatment
  Quality of life measured by the 3-level version of EQ-5D. Questions 1 to 3 (mobility)
  1 (no problem) to 3 (unable) Questions 4 to 6 (personal autonomy)
  1 (no problem) to 3 (unable) Questions 7 to 9 (current activities)
  1 (no problem) to 3 (unable) Questions 10 to 12 (pain/discomfort)
  1 (none) to 3 (extreme) Questions 13 to 15 (anxiety/depression)
  1 (none) to 3 (extreme) Question 16 (health status) Scale from 0 to 100 (worse health to better health)
Evaluation of quality of life | 12 months after treatment
  Quality of life measured by the 3-level version of EQ-5D. Questions 1 to 3 (mobility)
  1 (no problem) to 3 (unable) Questions 4 to 6 (personal autonomy)
  1 (no problem) to 3 (unable) Questions 7 to 9 (current activities)
  1 (no problem) to 3 (unable) Questions 10 to 12 (pain/discomfort)
  1 (none) to 3 (extreme) Questions 13 to 15 (anxiety/depression)
  1 (none) to 3 (extreme) Question 16 (health status) Scale from 0 to 100 (worse health to better health)
Evaluation of quality of life | 18 months after treatment
  Quality of life measured by the 3-level version of EQ-5D. Questions 1 to 3 (mobility)
  1 (no problem) to 3 (unable) Questions 4 to 6 (personal autonomy)
  1 (no problem) to 3 (unable) Questions 7 to 9 (current activities)
  1 (no problem) to 3 (unable) Questions 10 to 12 (pain/discomfort)
  1 (none) to 3 (extreme) Questions 13 to 15 (anxiety/depression)
  1 (none) to 3 (extreme) Question 16 (health status) Scale from 0 to 100 (worse health to better health)
Evaluation of quality of life | 24 months after treatment
  Quality of life measured by the 3-level version of EQ-5D. Questions 1 to 3 (mobility)
  1 (no problem) to 3 (unable) Questions 4 to 6 (personal autonomy)
  1 (no problem) to 3 (unable) Questions 7 to 9 (current activities)
  1 (no problem) to 3 (unable) Questions 10 to 12 (pain/discomfort)
  1 (none) to 3 (extreme) Questions 13 to 15 (anxiety/depression)
  1 (none) to 3 (extreme) Question 16 (health status) Scale from 0 to 100 (worse health to better health)
Evaluation of quality of life | 30 months after treatment
  Quality of life measured by the 3-level version of EQ-5D. Questions 1 to 3 (mobility)
  1 (no problem) to 3 (unable) Questions 4 to 6 (personal autonomy)
  1 (no problem) to 3 (unable) Questions 7 to 9 (current activities)
  1 (no problem) to 3 (unable) Questions 10 to 12 (pain/discomfort)
  1 (none) to 3 (extreme) Questions 13 to 15 (anxiety/depression)
  1 (none) to 3 (extreme) Question 16 (health status) Scale from 0 to 100 (worse health to better health)
The rate of patients in biochemical failure | 6 weeks after treatment
  The rate of patients in biochemical failure is measured by PSA dosage:
  * PSA > 0.2 ng for patients treated by radical surgery
  * PSA nadir +2 ng/mL (Phoenix criteria) for patients treated by HIFU
The rate of patients in biochemical failure | 3 months after treatment
  The rate of patients in biochemical failure is measured by PSA dosage:
  * PSA > 0.2 ng for patients treated by radical surgery
  * PSA nadir +2 ng/mL (Phoenix criteria) for patients treated by HIFU
The rate of patients in biochemical failure | 6 months after treatment
  The rate of patients in biochemical failure is measured by PSA dosage:
  * PSA > 0.2 ng for patients treated by radical surgery
  * PSA nadir +2 ng/mL (Phoenix criteria) for patients treated by HIFU
The rate of patients in biochemical failure | 12 months after treatment
  The rate of patients in biochemical failure is measured by PSA dosage:
  * PSA > 0.2 ng for patients treated by radical surgery
  * PSA nadir +2 ng/mL (Phoenix criteria) for patients treated by HIFU
The rate of patients in biochemical failure | 18 months after treatment
  The rate of patients in biochemical failure is measured by PSA dosage:
  * PSA > 0.2 ng for patients treated by radical surgery
  * PSA nadir +2 ng/mL (Phoenix criteria) for patients treated by HIFU
The rate of patients in biochemical failure | 24 months after treatment
  The rate of patients in biochemical failure is measured by PSA dosage:
  * PSA > 0.2 ng for patients treated by radical surgery
  * PSA nadir +2 ng/mL (Phoenix criteria) for patients treated by HIFU
The rate of patients in biochemical failure | 30 months after treatment
  The rate of patients in biochemical failure is measured by PSA dosage:
  * PSA > 0.2 ng for patients treated by radical surgery
  * PSA nadir +2 ng/mL (Phoenix criteria) for patients treated by HIFU
The rate of local recurrence | 3 months after treatment
  The rate of local recurrence is measured by control biopsy (number of positive biopsies)
Survival without metastases | 6 months after treatment
  demonstrated by an additional assessment (CT scan and bone scintigraphy, supplemented by MRI in case of suspicious anomaly), recorded on the date of diagnosis.
Survival without metastases | 12 months after treatment
  demonstrated by an additional assessment (CT scan and bone scintigraphy, supplemented by MRI in case of suspicious anomaly), recorded on the date of diagnosis.
Survival without metastases | 18 months after treatment
  demonstrated by an additional assessment (CT scan and bone scintigraphy, supplemented by MRI in case of suspicious anomaly), recorded on the date of diagnosis.
Survival without metastases | 24 months after treatment
  demonstrated by an additional assessment (CT scan and bone scintigraphy, supplemented by MRI in case of suspicious anomaly), recorded on the date of diagnosis.
Survival without metastases | 30 months after treatment
  demonstrated by an additional assessment (CT scan and bone scintigraphy, supplemented by MRI in case of suspicious anomaly), recorded on the date of diagnosis.

CONTACTS AND LOCATIONS:
Locations (49):
- France (48):
  - Centre Hospitalier d'Aix en Provence, Aix-en-Provence
  - Polyckinique du Beaujolais, Arnas
  - Clinique St Etienne, Bayonne
  - CHRU de Besançon, Besançon
  - Clinique St Vincent, Besançon
  - Clinique Tivoli-Ducos, Bordeaux
  - Clinique St Augustin, Bordeaux
  - CHU de Bordeaux, Bordeaux
  - Nouvelle clinique Bel Air, Bordeaux
  - CHR de Chambéry, Chambéry
  - Pôle Santé Léonard de Vinci, Chambray-lès-Tours
  - PôleSanté République, Clermont-Ferrand
  - Hôpitaux civils de Colmar, Colmar
  - Polyclinique du parc Drevon, Dijon
  - CHU de Dijon, Dijon
  - Cliniqe du Val d'Ouest, Écully
  - CHU de Grenoble, Grenoble
  - Hôpital Privé Drome Ardèche, Guilherand-Granges
  - Cliique du Pré, Le Mans
  - Clinique Bon Secours, Le Puy-en-Velay
  - CHRU de Lille, Lille
  - Clinique La Louvière, Lille
  - CHU de Limoges, Limoges
  - Hospices Civils de lyon, Lyon
  - Hôpital St Joseph, Marseille
  - AP-AM, Marseille
  - Clinique Beau Soleil, Montpellier
  - Clinique Diaconat-Roosevelt, Mulhouse
  - CHU de Nice, Nice
  - CHU de Nîmes, Nîmes
  - Fondation St Jean de Dieu - Clinique Oudinot, Paris
  - Clinique Turin, Paris
  - Hôpital St Joseph, Paris
  - Hôpital TENON, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Europeen Georges Pompidou, Paris
  - CH de pontoise, Pontoise
  - Clinique Courlancy, Reims
  - CHU de rennes, Rennes
  - Clinique Nantes Atlantis, Saint-Herblain
  - CH de Saintonge, Saintes
  - Clinique Rhéna, Strasbourg
  - Hôpital Foch, Suresnes
  - Clinique St Michel, Toulon
  - CHU de Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
  - Clinique St Jean du Languedoc, Toulouse
  - Clinique Océanne, Vannes
- CHU de guadeloupe, Pointe-à-Pitre, Guadeloupe

REFERENCES:
- [Derived] Ploussard G, Coloby P, Chevallier T, Occean BV, Houede N, Villers A, Rischmann P; HIFI group. Whole-gland or Subtotal High-intensity Focused Ultrasound Versus Radical Prostatectomy: The Prospective, Noninferiority, Nonrandomized HIFI Trial. Eur Urol. 2025 May;87(5):526-533. doi: 10.1016/j.eururo.2024.11.006. Epub 2024 Dec 4. PMID 39632125